CLINICAL TRIAL: NCT05950919
Title: Z 32201 - Effects of a Package of Evidence-based Interventions and Implementation Strategies Based on WHO PEN for People Living With HIV and Cardio-metabolic Conditions in Lusaka, Zambia: A Type II Hybrid Effectiveness-implementation Stepped Wedge Trial
Brief Title: Effects of a Package of Evidence-based Interventions and Implementation Strategies Based on WHO PEN for People Living With HIV and Cardio-metabolic Conditions in Lusaka, Zambia
Acronym: TASKPEN UH3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Centre for Infectious Disease Research in Zambia (Other); University of Zambia (Other); Ministry of Health, Zambia (Other Government); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-2252; 4UH3HL156389-03 (NIH)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: HIV; Non Communicable Diseases
Keywords: HIV; cardio-metabolic conditions; TASKPEN; Non Communicable Diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: hybrid effectiveness-implementation stepped wedge trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASKPEN (Experimental): The TASKPEN intervention is a package of five evidence-based intervention (EBI) components that enhances WHO's Package of Essential Noncommunicable Disease Intervention for Primary Care (WHO-PEN) and includes a multi-faceted implementation strategy centred on service integration within routine HIV care settings. The EBI components and multi-faceted strategy have been adapted to the Zambian setting during recently completed formative work."
  Interventions: Other: TASKPEN
- Standard of Care (No Intervention): Screening, diagnosis, and treatment of cardio-metabolic NCDs are generally unavailable in the clinical departments where most PLHIV seek and receive health services. When these services are available, they tend to be siloed and offered only for hypertension in general outpatient medical settings that provide urgent care-like services. Healthcare workers do not have protocolized algorithms for NCD management in HIV service delivery settings. NCD equipment is often unavailable in ART and differentiated service delivery (DSD) clinics; most health facilities do not offer haemoglobin A1c or lipid panel testing; and fragmented NCD supply chain management systems mean that essential medications for the management of hypertension, diabetes, and dyslipidemia are often unavailable

INTERVENTIONS:
Other: TASKPEN — The package of integrated HIV/NCD services:
  1. Integrated non-communicable/HIV care ("one stop shop" for services)
  2. WHO PEN protocols, algorithm, & training materials adapted for Zambia
  3. Access to cardio-metabolic condition screening & laboratory monitoring
  4. Non-communicable disease-focused electronic medical record module
  5. Strengthened NCD medication supply chain
  Arms: TASKPEN

SUMMARY:
The purpose of this study is to evaluate the effects of a multi-level intervention known as "TASKPEN," adapted from the World Health Organization (WHO) Package of Essential Noncommunicable Disease Interventions (WHO-PEN) for the Zambian public health system, on clinical and implementation outcomes for persons living with HIV (PLHIV) with co-morbid cardio-metabolic conditions in Lusaka, Zambia.

DETAILED DESCRIPTION:
This hybrid effectiveness-implementation stepped wedge trial will be used to evaluate the clinical effectiveness and implementation outcomes and strategies. Investigators will evaluate the effects of TASKPEN on the primary clinical effectiveness outcome of dual HIV/ cardio-metabolic non-communicable diseases (NCD) control at 12 months, and the secondary implementation outcome of intervention reach in the clinic population. Other secondary outcomes will include longitudinal changes in the Atherosclerotic Cardiovascular Disease (ASCVD) Risk Estimator, changes in quality of life per the WHOQOL-HIV-Bref, modification of grade III hypertension, and HIV viral suppression at different accepted thresholds (i.e., <1,000 c/mL, <200 c/ml, <50 c/ml). A cluster will be defined as one health facility and their associated catchment area population (i.e., together a study site). Sequential crossover of sites will take place, from control to intervention, until all 12 clusters (i.e., all 12 sites) are exposed to the intervention before the end of the study. Trained and experienced study staff will conduct a bio-behavioral survey at baseline with approximately 1,020 participants across all study sites before introduction of the TASKPEN intervention. After this baseline survey is completed, four randomly selected clusters (i.e., 4 facilities) will be switched to the TASKPEN intervention (the first orange shaded step in Figure 3) over a ~4-week introduction/ "wash out" period, and then continue with TASKPEN implementation until the end of the trial. Six months later, another survey with 1,020 participants who have not participated previously will be done across all 12 sites at time T1 right before a second block of two clusters (i.e., clusters 5 and 6) are switched to the TASKPEN intervention. After another 6 months, the survey will be repeated, this time as a midline survey, and another two clusters (i.e., clusters 7 and 8) will be switched to the TASKPEN intervention after survey completion. Six months later, at time T3, another survey will be completed with 1,020 participants who have not volunteered previously right before the final four randomly selected clusters (i.e., clusters 9 through 12) switch to the TASKPEN intervention. After all facilities/ sites have received the intervention for at least 6 months, a final "end-line survey" will be administered at time T4. Once the end-line survey is completed, a total of approximately 5,100 participants will have completed a survey.

To overcome the limitations inherent to cross-sectional assessments of patient outcomes, and to facilitate collection of more detailed longitudinal data, a "nested cohort," will be embedded in the larger trial reflecting a representative sample of approximately 320 survey participants with co-morbid cardio-metabolic NCDs identified through study surveys to carefully follow longitudinal clinical outcomes in PLHIV with these conditions.

Embedded in the trial will be concurrent mixed methods data collection to assess implementation outcomes and to understand the mechanisms by which the evidence-based intervention package and associated implementation strategies did, or did not, achieve their intended effects or acted through the conceptual model of change.

ELIGIBILITY:
Objective 1:

Cross-sectional patient surveys (n=5100): all HIV-infected adults aged 18 years and older who seek HIV services at the study sites.

Following the baseline survey, investigators will exclude anyone who previously participated in a study survey. Investigators will also exclude people who present for one time services or who plan to transfer their HIV care to another site. Finally, people unwilling or unable to provide written informed consent will be excluded.

For the nested cohort, inclusion (n=320) participants will need to have been enrolled in a study survey and have evidence of one or more of the following cardio-metabolic conditions or risk factors at the time of the survey:

* Any current tobacco use (any tobacco use within 30 days of the survey, whether daily or non-daily use);
* Hypertension as defined by WHO PEN/ HEARTS (i.e., systolic blood pressure (SBP) =140 mmHg and/or diastolic blood pressure (DBP) =90 mmHg);
* Diabetes mellitus as defined by WHO PEN/ HEARTS (i.e., random plasma glucose = 11.1 mmol/L, fasting plasma glucose = 7 mmol/L, and/or hemoglobin A1c = 48 mmol/mol or =6.5%; and/or compatible clinical diagnosis);
* Prediabetes (defined as having impaired fasting glucose of 6.1 to 6.9 mmol/L and/or haemoglobin A1c 42 to 48 mmol/mol or between 6.0-6.4%); and/or
* Dyslipidaemia (defined as total cholesterol =5.2 mmol/L or low-density lipoprotein =3.4 mmol/L).
* Investigators will exclude adults who have no documented evidence of HIV infection, or who do not have a cardio-metabolic NCD or risk factor of interest. Investigators will also exclude people who did not participate in a patient survey, plan to transfer their HIV care to another site, or are unwilling/ unable to provide written informed consent.

Objective 2 Participant inclusion criteria

In-depth interview (IDI) participants must be

* HIV-positive adults
* =18 years of age
* survey and/or cohort participants and
* had received HIV and/or NCD services at a TASKPEN study site.

Focus group discussion (FGD) participants must be:

* =18 years of age;
* a non-physician health care worker (NPHW) or community health worker (CHW)/ lay health provider involved with TASKPEN or integrated HIV/NCD service delivery; and
* generally familiar with HIV and/or NCD service delivery at their facility.

Key informant interview (KII) participants must be:

* =18 years of age;
* a facility-level ART, DSD, out-patient department (OPD), or relevant clinic leader/ manager/ in-charge, or policy maker at district, provincial, or national level in Zambia; and
* generally familiar with HIV and/or NCD-related issues in their community.

Implementation questionnaire participants must be:

* HIV-positive adults
* =18 years of age
* who had exposure to the TASKPEN intervention at a study site OR
* =18 years of age,
* a facility-level healthcare provider or manager at district, provincial, or national level in Zambia, and
* familiar with the TASKPEN intervention.

Costing study participants must be:

* HIV-positive adults
* =18 years of age
* who had received HIV and/or NCD services at a TASKPEN study site OR
* =18 years of age and
* a facility-level healthcare provider or manager at facility, district, provincial, or national level in Zambia, and generally familiar with HIV and/or NCD-related issues.

Participant exclusion criteria

* Investigators will exclude adult IDI participants who have no evidence of having received HIV and/or NCD services at the sites during the study period, adult implementation questionnaire
* participants who were not exposed/ familiar with the TASKPEN intervention, as well as - people unwilling or unable to provide written informed consent.
* Investigators will exclude any potential IDI, FGD, or KII study participant if they are unwilling or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5620 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants with both HIV Viral Suppression and Control of Hypertension, Diabetes and Tobacco Use | Month 12
  Dual control of HIV and cardio-metabolic NCDs is defined as: HIV RNA <1,000 copies/mL on most recent measure AND absence of the following: 1) uncontrolled systolic and diastolic hypertension; 2) uncontrolled diabetes mellitus; and 3) current tobacco smoking.
Number of Participants with both HIV Viral Suppression and Control of Hypertension, Diabetes and Tobacco Use | Month 12
  Dual control of HIV and cardio-metabolic NCDs is defined as: HIV RNA <1,000 copies/mL on most recent measure AND absence of the following: 1) uncontrolled systolic and diastolic hypertension; 2) uncontrolled diabetes mellitus; and 3) current tobacco smoking.

SECONDARY OUTCOMES:
Percent of Participants with Improvement in 10-year ASCVD Risk Score | up to 24 months
  Participants who experience numerical improvement in 10-year ASCVD risk score and experience improvement in risk category (for example, change from high risk to intermediate risk, high to borderline risk, borderline to low risk, etc.). Assessed at 12 and 24 months.
Change in Blood Pressure Control from Baseline to Month 12 | Baseline, Month 12
  Average numerical change in systolic and diastolic blood pressure.
Change in Blood Pressure Control from Baseline to Month 24 | Baseline, Month 24
  Average numerical change in systolic and diastolic blood pressure.
Number of Participants with Severe Hypertension | up to 24 months
  Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥120 mmHg. Assessed at Baseline, 12 and 24 months.
Percent of Participants with Severe Hypertension | 1, 12 and 24 months
  Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥120 mmHg
Average Change in Haemoglobin A1c and Fasting Glucose | Baseline up to 24 months
  Mean change in HgbA1c and/or fasting blood glucose from baseline at last assessment. Assessed at Baseline, 12 and 24 months.
Ideal Cardiovascular Health (CVH) | 1, 12, and 24 months
  Average change in Ideal CVH score on a 0-7 point Likert scale The Ideal CVH is based on the following factors: (1) Smoking: never or former smoker; (2) Body mass index<23 kg/m^2; (3) Physical activity: ≥150 min/wk of moderate-intensity physical activity, ≥75 min/wk of vigorous intensity physical activity, or ≥150 min/wk of moderate or vigorous intensity physical activity; (4) Diet: 4 or 5 healthy dietary components as defined below; (5) Total cholesterol <200 mg/dL; (6) Blood pressure <120/80 mm Hg; (7) Fasting glucose <100 mg/dL. For diet, the ideal metric is determined based on intake of fruits and vegetables (≥450 g/d), fish (≥198 g/wk), fiber-rich whole grains (≥85 g/d), sodium (<1500 mg/d), sugar-sweetened beverages (≤1 liter/wk).
  To calculate the ideal CVH score, each metric is given 1 point and the number of ideal CVH metrics is added up for each participant. The range of scores is 0 to 7 inclusive with higher scores indicating better cardiovascular health.
Number of Participants with HIV-1 Viral Suppression | 0, 12, and 24 months
  To be assessed at empirically supported thresholds of <1,000 c/mL, <200 c/mL, and <50 c/mL.
Percent of Participants with HIV-1 Viral Suppression | 0, 12, and 24 months
  To be assessed at empirically supported thresholds of <1,000 c/mL, <200 c/mL, and <50 c/mL.
Number of Participants Retained in HIV Care | 0, 12, and 24 months
  Number of participants with evidence of being retained in HIV care within the last ~180 days.
Percent of Participants Retained in HIV Care | 1, 12, and 24 months
  Percent of participants with evidence of being retained in HIV care within the last ~180 days.
Variation of Medication Possession Ratio (MPR) ART | 0, 12 and 24 months
  Number of days late for pharmacy refills by total days on treatment, and then subtracting that percentage from 100%--for antiretroviral therapy (ART).
Variation of Medication Possession Ratio (MPR) NCD Medications | 0, 12 and 24 months
  Number of days late for pharmacy refills by total days on treatment, and then subtracting that percentage from 100%--for NCD medications.
Number of Participants with an Increase in Quality of Life (QOL) | up to 24 months
  Number of participants with an increase in quality of life score. Assessed at 12 and 24 months.
  A version of the World Health Organization (WHO)QOL-HIV BREF will be used with 31 questions over 6 domains adapted to the Zambia context. We will present an overall score where a higher score indicate a higher quality of life. Most items are scaled in a positive direction, but some domains (i.e., #1, #2, #3, and #6) are scaled in a negative direction and will be recoded (as 6 minus question score) such that high scores reflect better quality of life. The mean score of items within each domain will be used to calculate a domain score. The means scores will then multiplied by 4 to make domain scores comparable with the overall scores used in the WHOQOL, so that scores range between 4 and 20. An overall average score across all 6 domains will be reported.
Percent of Participants with an Increase in Quality of Life | up to 24 months
  Percent of participants with an increase in quality of life score. Assessed at 12 and 24 months.
  A version of the WHOQOL-HIV BREF will be used with 31 questions over 6 domains adapted to the Zambia context. We will present an overall score where a higher score indicate a higher quality of life. Most items are scaled in a positive direction, but some domains (i.e., #1, #2, #3, and #6) are scaled in a negative direction and will be recoded (as 6 minus question score) such that high scores reflect better quality of life. The mean score of items within each domain will be used to calculate a domain score. The means scores will then multiplied by 4 to make domain scores comparable with the overall scores used in the WHOQOL, so that scores range between 4 and 20. An overall average score across all 6 domains will be reported.

OTHER OUTCOMES:
Number of Participants Reached | 0, 12, and 24 months
  Number of PLHIV at the clinic (i.e., with documented receipt of ART/ HIV care services at a study site) screened for hypertension at 0, 12, and 24 months from TASKPEN introduction
Percent of Participants Reached | 0, 12, and 24 months
  Percent of PLHIV at the clinic (i.e., with documented receipt of ART/ HIV care services at a study site) screened for hypertension at 0, 12, and 24 months from TASKPEN introduction
Number of Facilities Adopting TASKPEN | 0, 12, and 24 months
  Number of facilities and providers initiating TASKPEN intervention/ integrated care at 0, 12, and 24 months
Percent of Facilities Adopting TASKPEN | 0, 12, and 24 months
  Percent of facilities and providers initiating TASKPEN intervention/ integrated care at 0, 12, and 24 months
Level of Adherence to Implementation | 0, 12, and 24 months
  Percent of nurses and other non-physician health workers at each site that supported intervention/ integrated care implementation at least once at 0, 12 and 24 months
Mean Acceptability of Intervention Score | 6 months
  Average (mean) Acceptability of Intervention Measure (AIM) score after TASKPEN implementation at ≥6 months from TASKPEN introduction The "Acceptability of Intervention Measure (AIM)" is a 4-item instrument measuring the acceptability of an evidence-based practice or intervention. A scale can be created for this measure by averaging responses from each item.
  Scale values range from 1 (completely disagree) to 5 (completely agree). Higher scores indicate greater acceptability, feasibility, or appropriateness on the AIM, FIM, or IAM, respectively. No items need to be reverse coded.
Mean Feasibility of Intervention Score | 6 months
  Average (mean) Feasibility of Intervention Measure (FIM) score after TASKPEN implementation at ≥6 months from TASKPEN introduction The "Feasibility of Intervention Measure (FIM)" is a 4-item instrument measuring the feasibility of an evidence-based practice or intervention. A scale can be created for this measure by averaging responses from each item.
  Scale values range from 1 (completely disagree) to 5 (completely agree). Higher scores indicate greater acceptability, feasibility, or appropriateness on the AIM, FIM, or IAM, respectively. No items need to be reverse coded.
Mean Appropriateness of Intervention Score | 6 months
  Average (mean) Intervention Appropriateness Measure (IAM) score after TASKPEN implementation at ≥6 months from TASKPEN introduction The "Intervention Appropriateness Measure (IAM)" is a 4-item instrument measuring the appropriateness of an evidence-based practice or intervention. A scale can be created for this measure by averaging responses from each item.
  Scale values range from 1 (completely disagree) to 5 (completely agree). Higher scores indicate greater acceptability, feasibility, or appropriateness on the AIM, FIM, or IAM, respectively. No items need to be reverse coded.
Cost-effectiveness of intervention | 0, 12, and 24 months
  Incremental cost-effectiveness ratios (ICERs) at 0, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, MPH, Principal Investigator — University of North Carolina; Wilbroad Mutale, MBChB, MPhil, PhD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (12):
- Zambia (12):
  - Bauleni Health Center, Lusaka
  - Chawama 1st Level Hospital, Lusaka
  - Chelstone Urban Health Center, Lusaka
  - Chipata 1st Level Hospital, Lusaka
  - Kabwata Urban Health Center, Lusaka
  - Kalingalinga Urban Health Center, Lusaka
  - Kamwala Urban Health Center, Lusaka
  - Kanyama 1st Level Hospital, Lusaka
  - Makeni Urban Health Center, Lusaka
  - Mtendere Health Center, Lusaka
  - Ng'ombe Urban Health Center, Lusaka
  - Railway Urban Health Center, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Herce ME, Bosomprah S, Masiye F, Mweemba O, Edwards JK, Mandyata C, Siame M, Mwila C, Matenga T, Frimpong C, Mugala A, Mbewe P, Shankalala P, Sichone P, Kasenge B, Chunga L, Adams R, Banda B, Mwamba D, Nachalwe N, Agarwal M, Williams MJ, Tonwe V, Pry JM, Musheke M, Vinikoor M, Mutale W. Evaluating a multifaceted implementation strategy and package of evidence-based interventions based on WHO PEN for people living with HIV and cardiometabolic conditions in Lusaka, Zambia: protocol for the TASKPEN hybrid effectiveness-implementation stepped wedge cluster randomized trial. Implement Sci Commun. 2024 Jun 6;5(1):61. doi: 10.1186/s43058-024-00601-z. PMID 38844992